CLINICAL TRIAL: NCT01757002
Title: Pragmatic Randomized Controlled Trial of the Web-Based Asthma Management Intervention (Puff City) in Teens With Asthma Attending Urban Clinics
Brief Title: Web-Based and Tailored Asthma Management Intervention (Puff City) in Teens With Asthma Attending Urban Clinics
Acronym: PCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: University of Michigan (Other); Augusta University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dr. Mei Lu, Senior Biostatistician, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R01HL114981-01 (NIH); 1R01HL114981-01 (NIH)
Record Dates: First submitted 2012-12-07; First posted 2012-12-28 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: Urban adolescents; Acute asthma; Asthma; Computer tailoring; Web-based intervention; Puff City
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tailored asthma management program (Experimental): Teens randomized to the experimental arm will receive 4 sessions plus a booster of web-based, tailored asthma management.
  Interventions: Behavioral: Teens randomized to the experimental arm will receive 4 sessions plus a booster of web-based, tailored asthma management.
- Control (Active Comparator): Teens in the control group will receive generic, web-based asthma education.
  Interventions: Behavioral: Teens in the control group will receive generic, web-based asthma education.

INTERVENTIONS:
Behavioral: Teens randomized to the experimental arm will receive 4 sessions plus a booster of web-based, tailored asthma management. — Web-based, computer-tailored asthma management intervention delivered in 4 sessions, plus a 6 month booster.
  Arms: Tailored asthma management program
Behavioral: Teens in the control group will receive generic, web-based asthma education. — Web-based, generic asthma management intervention delivered in 4 sessions.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the Puff City web-based behavioral intervention of asthma management program in a clinical setting. This study also examines and evaluates the cost and efficiency of patient eligibility determination methods, patient recruitment, study monitoring (compliance with study regimen, participant retention and follow-up), and the collection of clinical endpoints.

DETAILED DESCRIPTION:
Asthma continues to be a major public health problem in the US with high economic and social costs. Vulnerable ethnic communities are disproportionately affected by asthma as demonstrated by higher morbidity and mortality for these groups. We have completed two school-based, randomized trials of a web-based, computer-tailored asthma management intervention that targets urban teens (Puff City).

The current study, Puff City in the Clinic, will be evaluated as a clinical tool by initiating the web-based behavioral intervention of asthma management in a clinical setting. However, the current paradigm for conducting such a trial is costly with respect to patient recruitment, intervention delivery, and data collection and management. To address these high costs, the study utilizes comparative effectiveness research (CER) pragmatic approaches to design a randomized controlled trial for patient recruitment and determination of eligibility, study monitoring (compliance with study regimen, participant retention and follow-up), and collection of clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

* 13-19 years of age
* Must be able to provide electronic assent and have consent from a parent/guardian if applicable
* Diagnosis of asthma by meeting one of the following criteria within the last 12 months:

  * At least one emergency department diagnosis of asthma or
  * At least one acute inpatient encounter with asthma as the principal diagnosis or
  * At least four outpatient visits with an asthma diagnosis and at least 2 asthma medications dispensed or
  * At least four asthma medications dispensed

Exclusion Criteria:

* Inability to provide informed consent/assent
* Lack of physician diagnosis of asthma
* Other co-morbidities that make it impossible for the individual to participate.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 266 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) | 12 Months
  Comparison of ACT scores at 12 months after the randomization

SECONDARY OUTCOMES:
Asthma Exacerbations/Functional Status | 12 Months
  Comparison of asthma exacerbations (asthma hospitalizations, emergency department visits, or oral corticosteroid dispensing)and functional status(e.g. self report of symptom-days, symptom nights, days of restricted activity, school/work days missed) at 12 months after randomization.

OTHER OUTCOMES:
The Cost | Up to 12 months
  The cost of study intervention will be evaluated: The cost for participant enrollment with Electronic Medical Record (EMR) initiation; data collection and management with/o EMR initiation including assessing the reliability of EMR clinical outcomes/primary endpoints, compared to chart abstraction.
The Cost Effectiveness | Up to 12 months
  The cost effectiveness of Puff City intervention compared to controls without study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Lu, PhD, Principal Investigator — Henry Ford Health System; Christine Joseph, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Derived] Lu M, Ownby DR, Zoratti E, Roblin D, Johnson D, Johnson CC, Joseph CL. Improving efficiency and reducing costs: Design of an adaptive, seamless, and enriched pragmatic efficacy trial of an online asthma management program. Contemp Clin Trials. 2014 May;38(1):19-27. doi: 10.1016/j.cct.2014.02.008. Epub 2014 Mar 6. PMID 24607295